CLINICAL TRIAL: NCT02071459
Title: Evaluate the Long-term (3 Months) Efficacy of L-threo DOPS (DroxiDopa) on Orthostatic Hypotension Symptoms and Other Non-motor Symptoms in Patients With Multiple System Atrophy (MSA). Comparative Study Versus Placebo
Brief Title: Efficacy of L-threo DOPS on Orthostatic Hypotension Symptoms and Other Non-motor Symptoms in Patients With MSA
Acronym: DOPS-AMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12 554 01; 12-018-0200 (Other Grant/Funding Number: French Ministry of Health, PHRC 2012)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Multiple System Atrophy
Keywords: L-threo DOPS (DroxiDopa); Orthostatic Hypotension; Multiple system atrophy
MeSH Terms: conditions — Multiple System Atrophy; Hypotension, Orthostatic | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Threo DOPS (Experimental): patients with Multiple System Atrophy (MSA) after 12 weeks to continued therapy with L-Threo DOPS
  Interventions: Drug: L-Threo DOPS
- placebo (Placebo Comparator): patients with Multiple System Atrophy (MSA) after 12 weeks to continued therapy with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L-Threo DOPS — initial dose titration period (4 weeks) followed by 8 weeks at the max tolerated dose
  Other Names: L DOPS or DroxiDopa
  Arms: L-Threo DOPS
Drug: placebo — initial period (4 weeks) followed by 8 weeks
  Arms: placebo

SUMMARY:
Evaluate the effects of L-Threo DOPS on orthostatic hypotension symptoms and other non-motor symptoms in patients with Multiple System Atrophy (MSA) after 12 weeks following randomization to continued therapy with droxidopa or placebo.

DETAILED DESCRIPTION:
Background :

Multiple system atrophy (MSA) is a rare, sporadic progressive neurodegenerative disorder, rapidly leading to severe disability and impairment of quality of life. MSA is characterized by a variable combination of a poor levodopa parkinsonism and /or cerebellar ataxia and autonomic failure (cardiovascular and / or bladder and sexual dysfunction) (Gilman et al, 2008). The prevalence is approximately 4-5 cases per 100 000 inhabitants.

Orthostatic hypotension (OH) is one of the major symptoms of MSA, present in a large majority of patients, leading to significant disability because of impaired balance, falls and possibly syncope. Drugs available to treat OH in this disease are very limited.

L-ThreoDOPS (L DOPS or DroxiDopa) is an orally administered synthetic catecholamine acid that is converted to the sympathetic neurotransmitter norepinephrine (NE) through a single step of decarboxylation by the endogenous enzyme 3,4-dihydroxyphenylalanine (DOPA) decarboxylase. It prevents symptoms related to OH by central and/peripheral mechanisms. This drug is currently developed for "neurogenic OH" by Chelsea Therapeutics on the basis of short duration placebo-controlled randomized trials. Besides an expected effect on OH, L-DOPS may also, by noradrenergic stimulation, improve some motor and non-motor symptoms common and disabling in MSA patients such as akinesia and fatigue.

In this context, the French reference center for MSA and the 12 national centers with identified skills to manage this disease, propose to conduct a national multicenter randomized clinical trial versus placebo to evaluate the long term efficacy (3 months) of L-threo DOPS on the OH and other non-motor symptoms in MSA patients.

ELIGIBILITY:
Inclusion Criteria:

* MSA patients (possible or probable, MSA-P or C (according to revised criteria, Gilman et al 2008)).
* Aged 30 to 80 years,
* Able to walk at least 10 meters
* With symptomatic OH (score of at least 3 at one of the items of Part I of the OH scale (OHQ))
* Documented fall in systolic blood pressure of at least 20 mmHg, and/or in diastolic blood pressure of at least 10 mmHg, within 3 minutes after standing.
* Able to fill in the evaluation questionnaires with or without help
* With no significant problems with swallowing.
* Stable anti-parkinsonian, dysautonomia and depression treatments for the 4 weeks before the study and during the entire study
* Signed written informed consent for the present study.

Exclusion Criteria:

* Dementia (DSM-IV, Mini-Mental State Examination (MMSE) < 24/30)
* Concomitant use of vaso-constrictive drugs, other than midodrine. Patients taking vasoconstrictor agents such as ephedrine, dihydroergotamine, must stop taking these drugs at least 2 days or 7 half-lives prior to their baseline visit (Visit 1); the association with midodrine may be kept at a stable dose not exceeding 3 tablets (7.5 mg) / day if the patient has no CV history. This will be discussed case by case with the coordinating center and the safety committee of this study.
* Taking anti-hypertensive medication

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of long term efficacy of L-threo DOPS | 12 weeks
  Evaluate the efficacy of long term efficacy of L-threo DOPS (droxidopa) in MSA patients (probable or possible - cerebellar (C) or parkinsonian (P) type) with symptomatic NOH as measured by the relative change in mean score of Orthostatic Hypotension Symptom Assessment (OHSA) (Part I of the questionnaire on the symptoms OH (OHQ) (Kaufmann et al., 2011)) 12 weeks following randomization to therapy with droxidopa or placebo (including 8 weeks to maximum tolerated dose).

SECONDARY OUTCOMES:
efficacy of L-ThreoDOPS on symptomatic OH | 12 weeks
  Evaluate and compare the efficacy of L-ThreoDOPS on symptomatic OH (measured by the relative change in mean score of Item 1 of the Orthostatic Hypotension Symptom Assessment (OHSA)) in MSA patients 4, 8 and 12 weeks following randomization to continued therapy with droxidopa or placebo
effects of L-Threo DOPS on motor symptoms | 12 weeks
  Evaluate the effects of L-Threo DOPS on motor symptoms (UMSARS I and II) in MSA patients after 12 weeks following randomization to continued therapy with droxidopa or placebo
effect of L-Threo DOPS on dysautonomic symptoms | 12 weeks
  Evaluate the effect of L-Threo DOPS on dysautonomic symptoms (COMPASS) in MSA patients after 4, 8 and 12 weeks following randomization to continued therapy with droxidopa or placebo
safety of high doses of L-ThreoDOPS | 12 Weeks
  Determine the safety of high doses of L-ThreoDOPS in MSA patients based on the occurrence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Anne PAVY-LE-TRAON, PHD, Principal Investigator — University Hospital, Toulouse
Locations (13):
- France (13):
  - Centre hospitalier d'Angers, Angers
  - CHU bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHRU de lille, Lille
  - CHU de limoges, Limoges
  - Hôpital La Timone, Marseille
  - Hôpital G. & R. Laennec, Nantes
  - Hôpital Pitié-Salpétrière, Paris
  - CHU de Poitiers, Poitiers
  - CHU Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - chu de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No